CLINICAL TRIAL: NCT03078920
Title: Subjective and Objective Benefits of a Contralateral Routing of Signals (CROS) System in Unilateral Cochlear Implant Recipients
Brief Title: Benefits of a Contralateral Routing of Signals (CROS) System in Unilateral CI-recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ABIntl-16-04
Record Dates: First submitted 2017-02-21; First posted 2017-03-14 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 11 unilateral adult cochlear implant users (Other): Speech Reception Threshold (SRT) measured with an adaptive test
  Interventions: Device: Naída CROS

INTERVENTIONS:
Device: Naída CROS — At fitting Naída CROS and a loaner Naída CI processor are used for the duration of the study. The fitting software allows to enable a HIBAN link between the CI processor and the Naída CROS. The fitting of the CI processor is based on the clinical programming of the subject. No changes are made to the fitting parameters unless the subject requests changes. The fitting is done according to the clinical routine. The Naída CROS is pre-configured to communicate with the Naída CI when switched on.

SUMMARY:
The objective is to investigate the new Naida CROS device in adult recipients including chronic phases and to generate some preliminary pre-launch data.

The formal study objectives are to compare the speech intelligibility in quiet and noise when using the CROS device with the Naida CI Q70 processor versus the Naida CI processor alone in quiet and noise conditions. Subjects will be tested with and without CROS at the baseline visit and then at follow-up visits taking place one month and three months after baseline. Subjects will use the new device at home between the first two visits appointments and then will only use the Naida CI processor for two additional weeks to better evaluate the handicap of not having access to contralateral signal input. There will be four visits to the centre in total.

Subjective feedback will be collected through questionnaire like the APHAB and Speech, Spatial and Qualities of Hearing Scale (SSQ). A customised questionnaire focusing usability and benefit of the CROS will also be administered.

Additional interest of the study will be to evaluate any acclimatisation effect with the CROS device both objectively and subjectively.

DETAILED DESCRIPTION:
Nowadays, cochlear implants (CI) are widely used prostheses for deaf people. They are stimulating the auditory nerve cells electrically, circumventing the tympanic membrane and ossicles of the middle ear and the inner and outer hair cells of the inner ear. A single cochlear implant usually provides substantial benefit to recipients who were previously severe-to-profoundly deaf. In quiet listening situations, scores for the perception of sentences typically show a strong ceiling effect . However, in even moderately challenging listening situations, where speech needs to be understood when presented at lower levels or in the presence of competing noise, speech perception scores drop to below the level required to support practical communication. The speech reception threshold (SRT), the signal-to-noise ratio (SNR) required to understand 50% of words in sentences for normal hearing subjects listening in their first language, is around -6 decibel (dB). For CI recipients this can be +9 to +15 dB. These figures relate to a test situation where target speech comes from directly in front of the CI recipient. If sound comes from their un-implanted side, it will typically suffer a further 6 dB of attenuation, a figure in agreement with published literature, with the information rich higher frequencies being even more attenuated. This puts unilaterally implanted CI users in a very difficult position. Bilateral cochlear implantation has been shown to provide advantages although its main advantage is in dealing with the head shadow problem, rather than restoring true binaural hearing advantages such as spatial release from masking. Bilateral implantation is obviously expensive and not available to adults in many countries. In addition, some subjects cannot get a second implant due to medical reasons or they do not want to undergo a second surgery. These subjects will have similar limitations as single-sided deaf (SSD) patients: due to the head shadow effect, soft sounds from the direction of the non-implanted side will not be heard. To overcome these limitations, the contralateral routing of signals (CROS) by means of a contralateral receiver could be a very beneficial tool. This system has already been used in the hearing instrument field for a while and showed benefit to patients suffering from single-sided deafness. Some preliminary studies using experimental devices were also conducted with cochlear implants users showing similar benefits.

A comparable system, the Naída CROS device, developed by Advanced Bionics as contralateral receiver will be evaluated in this study. The Naída CROS device is placed on the contralateral ear similar to a small hearing aid. It captures the incoming sound and transmits it wirelessly to the CI sound processor. In the sound processor, signals from both the ipsilateral and the contralateral side are mixed together.

While some work has been done acutely with hearing instrument prototypes, this study will evaluate the Naída CI device with the Naída CROS device and involve take home experience. The study will evaluate the benefit of adding a CROS device to unilaterally implanted subjects both objectively and subjectively.

A microphone is placed at the unilateral CI recipient's non-implanted ear. This microphone can then detect sounds from the head-shadowed side and route them to the CI sound processor. In the hearing instrument field such systems have been commonly applied for cases of unilateral deafness and are referred to as contralateral routing of signal or CROS systems. The most recent Advanced Bionics sound processors, the Naída CI Q70 and Q90, have the ability to communicate wirelessly with another Naída CI processor, or with some Phonak hearing instrument models, including a CROS device, placed on the contralateral ear. The full microphone signal is transmitted wirelessly to the Naída CI sound processor and can be mixed with the microphone signal from the implanted side. The Naída CROS device is based on the Phonak CROS H20 device hardware. It contains essentially a microphone, radio transmitter and battery so it is small and discrete. The Naída CROS device is designed to be an out-of-the-box solution to work automatically with the Naída CI without the need for fitting.

The Naída CI processors will be programmed using the conventional fitting software SoundWave (version 3.1) provided by Advanced Bionics, to enable wireless communication between the CI and Naída CROS devices. The software is not yet CE approved, but is tested with respect to the company's internal standards. The CE approved CI system as a whole is still used in its intended way during the study, i.e. to "restore a level of auditory sensation". All basic safety features incorporated in the implant system remain active and are not affected by the study. The Naída CROS device also works in its intended way without the need for programming. However, the investigational Naída CROS device will be pre-configured with a research software to instantaneously communicate with the approved Naída CI processor when switched on.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Unilaterally implanted with an Advanced Bionics Clarion or HiRes90k (implant type) implant
* At least 6 months of cochlear implant use
* At least 3 months experience with the Naída CI processor
* No benefit or limited benefit with a contralateral hearing aid
* Minimum speech understanding level in quiet of 30% (Lafon lists)
* Ability to wear the Naída CROS device on their contralateral ear and to have sufficient dexterity and understanding to handle both the Naída CI and CROS devices
* Able to describe the sound quality that they receive
* French language proficiency

Exclusion Criteria:

* Persons mentioned in the following articles of the French public health code: articles from L. 1121-5 to L.1121-8
* Participating in another clinical study
* Difficulties additional to hearing impairment that would interfere with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Speech Reception Threshold (SRT) measured with an adaptive test (French Matrix sentence test) | Baseline
  Speech tests in quiet & noise with the Naída CI processor alone and with the Naída CROS device
Speech Reception Threshold (SRT) measured with an adaptive test (French Matrix sentence test) | 1 month
  Speech tests in quiet & noise with the Naída CI processor alone and with the Naída CROS device
Speech Reception Threshold (SRT) measured with an adaptive test (French Matrix sentence test) | 3 months
  Speech tests in quiet & noise with the Naída CI processor alone and with the Naída CROS device
Speech Reception Threshold (SRT) measured with an adaptive test (French Matrix sentence test) | Baseline
  Questionnaires about Naída CI sound processor and Naída CROS device listening condition
Speech Reception Threshold (SRT) measured with an adaptive test (French Matrix sentence test) | 1 month
  Questionnaires about Naída CI sound processor and Naída CROS device listening condition
Speech Reception Threshold (SRT) measured with an adaptive test (French Matrix sentence test) | 3 months
  Questionnaires about Naída CI sound processor and Naída CROS device listening condition

SECONDARY OUTCOMES:
Questionnaires about Naída CI sound processor listening condition | Baseline
  Evaluate the benefit/usability of the Naída CROS device in everyday life
Questionnaires about Naída CI sound processor listening condition | Baseline
  Evaluate any acclimatization effect of using the Naída CROS device
Questionnaires about Naída CI sound processor listening condition | 1 months
  Evaluate the benefit/usability of the Naída CROS device in everyday life
  • Evaluate any acclimatization effect of using the Naída CROS device
Questionnaires about Naída CI sound processor listening condition | 1 months
  Evaluate any acclimatization effect of using the Naída CROS device
Questionnaires about Naída CI sound processor listening condition | 3 months
  Evaluate the benefit/usability of the Naída CROS device in everyday life
Questionnaires about Naída CI sound processor listening condition | 3 months
  Evaluate any acclimatization effect of using the Naída CROS device
Questionnaires about Naída CI sound processor listening condition | 3.5 months
  Evaluate the benefit/usability of the Naída CROS device in everyday life
Questionnaires about Naída CI sound processor listening condition | 3.5 months
  Evaluate any acclimatization effect of using the Naída CROS device

CONTACTS AND LOCATIONS:
Overall Officials: Volkmar Hamacher, Dr., Study Chair — Advanced Bionics GmbH; Isabelle MOSNIER, Dr., Principal Investigator — Groupe Hospitalier de la PITIE-SALPETRIERE
Locations (1):
- Groupe Hospitalier de la PITIE-SALPETRIERE, Paris, France

IPD SHARING:
Plan to Share IPD: No